CLINICAL TRIAL: NCT05024773
Title: A Phase III, Single-arm Study to Evaluate the Efficacy and Safety of ONCOFID-P-B (Paclitaxel-hyaluronic Acid Conjugate) Administered Intravesically to Patients With BCG-unresponsive Carcinoma in Situ of the Bladder With or Without Ta-T1 Papillary Disease (Orion-BC)
Brief Title: Study of ONCOFID-P-B (PACLITAXEL-HYALURONIC ACID)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R39_21_01
Record Dates: First submitted 2021-08-20; First posted 2021-08-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Bladder Carcinoma in Situ (CIS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ONCOFID P-B (PACLITAXEL-HYALURONIC ACID) (Experimental)
  Interventions: Drug: ONCOFID P-B (PACLITAXEL-HYALURONIC ACID)

INTERVENTIONS:
Drug: ONCOFID P-B (PACLITAXEL-HYALURONIC ACID) — Schedule: once a week for 12 consecutive weeks (induction phase). Patients who achieve a complete response at the end of the induction phase will enter the maintenance phase, during which ONCOFID-P-B is administered once a month for 12 months until recurrence or progression of the disease.

SUMMARY:
This is a phase III, single-arm, multicenter, international study to assess the efficacy and safety of ONCOFID-P-B following intravesical instillation in adult patients with histologically and cytologically confirmed CIS, with or without concomitant Ta-T1, who are unresponsive to BCG therapy and unwilling or unfit to undergo radical cystectomy.

After providing written informed consent (in presence of an Independent Witness, if applicable), patients will receive an induction therapy consisting of 12 weekly intravesical instillations of ONCOFID-P-B (induction phase). Patients with residual CIS at the end of induction treatment are eligible to enter a re-induction course of therapy (reinduction phase). Patients with stable disease by Investigator assessment defined as neither increased or decreased in extent or severity compared to baseline, are not eligible for re-induction therapy. Patients who achieve a complete resonde (CR) at the end of the induction or re-induction phase enter in the maintenance phase and receive monthly intravesical instillations of ONCOFID-P-B for an additional 12 monsthe or untile recurrence of CIS/HG Ta-T1 or progression to MIBC or extravesical disease. Patients who do not achieve a CR at the end of induction or re-induction phase, will discontinue investigational treatement and are followed up until month 48 from induction or re-induction start, or until a new antitumor therapy is initiated, wichever occurs first.

Tumor response is evaluated by cystoscopy, cytology and biopsy at the end of the induction and re-induction phases and at Safety Follow Up Visit (SFUV). During the maintenance/follow-up period, tumorresponse is evaluated by cystoscopy and cytology every 3 months for up to 24 months from induction or re-induction start, and then every 6 months for an additional 2 years (long-term follow-up). Tumor biopsies are performed in case of of positive cystoscopy and/or cytology. Random biopsies are to be performed at 6, 12 and 18 months after the end of the induction or re-induction phase in responding patients (i.e. at 9, 15 and 21 months after induction or re-induction start.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to freely provide written informed consent (in presence of an Independent Witness if applicable) prior to performing study procedures.
2. Age 18 years or older, male or female.
3. Persistent or recurrent histologically confirmed CIS of the bladder with or without concomitant recurrent HG Ta-T1 and with no evidence of metastases demonstrated by abdominal CT scan or MRI.
4. "BCG unresponsive" patients who refuse radical cystectomy or are not clinically suitable for cystectomy. BCG unresponsive disease is defined as persistent or recurrent CIS alone or with recurrent HG Ta-T1 within 12 months of completion of adequate BCG therapy.

   Adequate BCG therapy is defined as at least one of the following:
   * At least five of six doses of an initial induction course plus at least two of three doses of maintenance therapy.
   * At least five of six doses of an initial induction course plus at least two of six doses of a second induction course.
5. Complete resection of Ta-T1 papillary lesions before entering the trial in patients with concomitant CIS and papillary tumors (residual CIS acceptable, obvious areas of CIS should also be fulgurated).

   1. In patients with T1 papillary lesions undergoing resection of the base of the lesion, the biopsy should contain muscle fibers.
   2. In patients undergoing transurethal resection of their bladder tumors, absence of locally advanced disease should be confirmed by pelvic examination under anesthesia.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
7. Adequate organ function:

   * absolute neutrophil count ≥ 1,500/mm3,
   * platelets ≥ 100,000/mm3,
   * hemoglobin ≥ 8.5 g/dL,
   * ALT/AST ≤1. 5 x upper limit of normal (ULN),
   * alkaline phosphatase ≤ 5 x ULN,
   * total serum bilirubin ≤ 1.5 x ULN, for patients with Gilbert's ≤ 3 X ULN,
   * serum creatinine ≤ 2.2 mg/dL.
8. Women in non-reproductive years (defined as surgically sterile or one year postmenopausal). Women of childbearing potential (WOCBP) must have a negative serum pregnancy test upon entry into this study and agree to use highly effective contraceptive methods, i.e. methods that can achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include:

   * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

     * oral
     * intravaginal
     * transdermal
   * progestogen-only hormonal contraception associated with inhibition of ovulation:

     * oral
     * injectable
     * implantable
   * intrauterine device (IUD)
   * intrauterine hormone-releasing system (IUS)
   * bilateral tubal occlusion
   * vasectomised partner (*)
   * sexual abstinence (**)
9. Male patients with WOCBP partners must agree to use effective contraceptive methods, i.e.:

   * condom;
   * consider contraception for non-pregnant WOCBP partner.
10. Able and willing to comply with the scheduled visits, therapy plans, and laboratory tests required in this protocol.

(*) Vasectomised partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomised partner has received medical assessment of the surgical success.

(**) Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated to the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

Exclusion Criteria:

1. Current or previous muscle-invasive disease (T2-T4) or metastatic urothelial carcinoma.
2. Patients with more than 12 months between inclusion and the last BCG instillation
3. Suspected hypersensitivity to paclitaxel or to any of the Oncofid-P-B constituents.
4. Previous or concomitant cancer of the upper urinary tract or the prostatic urethra. Freedom from upper tract disease must be demonstrated by intravenous pyelogram, retrograde pyelogram, CT scan or MRI.
5. Current or prior systemic therapy for bladder cancer.
6. Intravesical therapy within 4 weeks prior to beginning study treatment with the exception of cytotoxic agents (e.g. mitomycin C, doxorubicin and epirubicin) when administered as a single instillation immediately following a TURBT procedure between 14 to 60 days prior to beginning study treatment.
7. Symptomatic urinary tract infection or bacterial cystitis. Once successfully treated (negative urine culture), patients may enter the study.
8. Major surgery, other than diagnostic, within 4 weeks prior to treatment.
9. Patients who have previous or concurrent malignancies that require treatment and are not clinically stable; examples of permitted concurrent recent second malignancies are: adequately treated basal cell or squamous cell skin cancer, in situ carcinoma of the cervix or prostate cancer on active surveillance at low risk for progression, defined as prostate-specific antigen (PSA) <10 ng/dL, Gleason score 6 or less and cT1.
10. Subjects who, in the opinion of the Investigator, cannot tolerate intravesical administration or intravesical surgical manipulation (cystoscopy, biopsy) due to the presence of serious comorbid condition(s) (e.g., uncontrolled cardiac or respiratory disorders).
11. Presence of significant urologic disease interfering with intravesical therapy.
12. Current enrollment or participation in another therapeutic clinical trial within 6 months preceding screening. Patients previously included in a BCG-only study arm might be enrolled following discussion with the medical monitor and/or sponsor if the definition of adequate BCG therapy is met.
13. Known substance and/or alcohol abuse.
14. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry in this study or could compromise protocol objectives.
15. Pregnancy, lactating women or women of childbearing potential (WOCBP) unwilling to use adequate birth control measures for the duration of the study and until 3 months after the end of treatment.
16. Male patients with WOCBP partners unwilling to use contraceptive methods for the duration of the study and until 6 months after the end of treatment.
17. Subjects who have a mean QTc >480 msec at baseline and who need concomitant medications which may cause QT prolongation.

    Applies to France Only:
18. Persons deprived of liberty by judical or administrative decision, adults subjects to a legal protection measure (under guardianship/curators), persons under protective measures and persons not affiliated with social security will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Centrally assessed Complete Response Rate (CRR) at any time | CRR will be evaluated at any time
  CRR calculated as the proportion of patients achieving a CR at any time. CRR will be based on central assessment of response

SECONDARY OUTCOMES:
Centrally assessed CRR | CRR will be evaluated at 6, 9, 12, 15, 18, 21, 24, 30, 36, 42 and 48 months after induction or re-induction
  CRR calculated as the proportion of patients achieving a CR at 6, 9, 12, 15, 18, 21, 24, 30, 36, 42 and 48 months after induction or re-induction start
Duration of Response (DoR) | DoR will be evaluated at 6, 9, 12, 15, 18, 21, 24, 30, 36, 42 and 48 months after induction or re-inductiononths after treatment start
  DoR defined as the time from first documented evidence of CR to time of documented recurrence (CIS or Ta-T1), progression to MIBC, to extravesical disease, or death
Duration of Response (DoR) rate | DoR rates will be evaluated at 6, 9, 12, 15, 18, 21, 30, 36, 42 and 48 after induction or re-induction start
  DoR rate calculated as the proportion of patients who maintained a CR after 6, 9, 12, 15, 18, 21, 30, 36, 42 and 48 months after induction or re-induction start.
Progression rate | Progression rate will be evaluated at EOIT/EROIT, 15, 24 and 48 months after induction or re-inductionstart
  Progression rate calculated as the proportion of patients with muscle invasion or extravesical expansion of the disease at EOIT/EORIT, 15, 24 and 48 months after induction or re-induction start
Time to progression | Time to progression will be evaluated at 15, 24 and 48 months after induction or re-induction start
  Time to progression defined as time from treatment start to time of documented tumor progression to MIBC or extravesical disease.
Rate of patients undergoing cystectomy | Rate of patients undergoing cystectomy will be evaluated at EOIT/EROIT, 9, 15, 24, 24 and 48 months after induction or re-induction start.
  Proportion of patients undergoing cystectomy for disease progression at EOIT/EORIT, 9, 15, 24 and 48 months after induction or re-induction start.
Time to cystectomy defined as time from start of treatment to the date of cystectomy | from start of treatment to date of cystectomy
  Time to cystectomy is defined as the time (months) form start of treatment to the date of cystectomy, analyzed using the Kaplan-Meier method. The median time to cystectomy will be presented along with 95% CI.
event-free survival (EFS) | Event-free survival (EFS) will be evaluated at any time during the study up to 48 months after treatment start
  EFS defined as time from treatment start to the time of documented recurrence after CR, or progression or death due to any cause.
Overall survival (OS) | overall survival (OS) will be evaluated at any time during the study up to 48 months after treatment start
  OS defined as time from treatment start to death due to any cause.
Incidence of Treatment-Emergent Adverse Events (Overall Safety) | Safety data will be evaluated up to study month 16
  Overall safety and tolerability evaluated throughout the study on the basis of the incidence, nature, severity and causality of TEAEs, coded to preferred term and system organ class (SOC) using the Medical Dictionary for Regulatory Activities (MedDRA) and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5 and the incidence of serious adverse events (SAEs)
Treatment time of retention (tolerability) | Tolerability will be evaluated up to study month 16
  The tolerability of ONCOFID-P-B expressed as the ability to retain intravesical instillation for the desired dwell time (optimal retention time is 120 minutes) and measured as time of retention.

CONTACTS AND LOCATIONS:
Locations (47):
- United States (6):
  - Banner Health- MD Anderson Cancer Center, Gilbert, Arizona
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - TriState Urologic Services PSC Inc. dba The Urology Group, Cincinnati, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
- France (7):
  - CHU Bordeaux -Hopital Pellegrin, Bordeaux
  - CHU de Clermont-Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU de Lille - Hopital Claude Huriez, Lille
  - Institute Paoli-Calmettes, Marseille
  - AP-HP Hopital Bichat-Claude Bernard, Paris
  - AP-HP Hopital Tenon, Paris
  - Centre Hospitalier Universitaire Poitiers, Poitiers
- Italy (12):
  - Humanitas Gavazzeni, Bergamo
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - Istituto Oncologico Veneto-I.R.C.C.S.-Ospedale San Giacomo, Castelfranco Veneto
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - ASL Lecce- Ospedale Vito Fazzi, Lecce
  - Istituto Clinico Humanitas, Milan
  - IRCSS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - IFO-Istituto Nazionale dei Tumori Regina Elena, Roma
  - AOU Città della Salute e della Scienza di Torino-Ospedale le Molinette, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona-Ospedale Borgo Trento, Verona
- Poland (3):
  - Wojewodzki Szpital im Sw. Ojca Pio w Przemyslu, Oddzial Urologiczny z Pododdzialem Urologii Onkologicznej, Przemyśl, Poland
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. prof. dr hab. med. Eleonory Reicher, Warsaw, Warszawa
  - Centrum Onkologii Ziemi Lubelskiej im. sw. Jana z Dukli, Oddzial Urologiczny, Lublin
- Spain (12):
  - Vall d'Hebron Barcelona Hospital, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona, Barcelona
  - Instituto Valenciano de Oncologia, Valencia, Valencia
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Fundación Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
- United Kingdom (7):
  - Darent Valley Hospital, Dartford, Kent
  - Huddersfield Royal Infirmary, Huddersfield
  - St James's University Hospital, Leeds
  - Barts Health NHS Trust, London
  - Derriford Hospital, Plymouth
  - Royal Preston Hospital, Preston
  - Royal Marsden Hospital - Surrey, Sutton